CLINICAL TRIAL: NCT03959930
Title: Transdermal Fluid Removal in Fluid Overload
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: British Heart Foundation (Other); Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B00097
Record Dates: First submitted 2019-04-17; First posted 2019-05-22 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Heart Failure; Odema
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional arm (Experimental): Total and segmental body fluid volumes (total water, extracellular water and interstitial water) will be measured by Segmental Bioelectrical Impedance Spectroscopy (as per manufacturer instructions of use). Areas with most significant oedema and skin in a suitable condition shall be selected for the TFR application. Moisture Meter shall be used at the selected site to measure the skin water content at 4 depths (0.5mm, 1.5mm, 2.5mm and 5mm).
  Interventions: Device: Transdermal Fluid Removal

INTERVENTIONS:
Device: Transdermal Fluid Removal — The Transdermal Fluid Removal (TFR) device is designed for use on the lower limbs of patients with Chronic Heart Failure and treatment resistant peripheral oedema.
  The TFR device is intended to be applied on oedematous skin of eligible patients, for periods of up to 10 hours at a time, to gently remove excess fluid through the skin, over a period of a few days during exacerbations, thereby avoiding hospitalisation for intravenous diuretics.
  The TFR device is designed to be used in conjunction with standard Negative Pressure Wound Therapy (NPWT) devices which are currently CE Marked and approved for use in both acute and homecare environment.
  Other Names: TFR

SUMMARY:
The proposed study seeks to explore the possibility of significantly increasing the success rate (from the current rate of 28%) of clinically significant Transdermal Fluid Removal (TFR) in heart failure patients. It seeks to further understand the device and patient characteristics influencing successful clinically relevant fluid removal and to measure any patient-defined benefits. It also wishes to explore the patient experience of the removal.

DETAILED DESCRIPTION:
Fluid overload is distressing and is particularly prevalent in patients with vital organ dysfunction such as in kidney and heart disease. Due to the patient's inability to remove excess wastes and water, these accumulate in their body fluid compartments. Such excess fluid and toxins have to be removed with high dose diuretics (water tablets or injections) or by frequent dialysis. Treatment with diuretics is effective initially in some patients but is fraught with risks and side effects. The retained fluid and wastes are mainly lodged within the extracellular compartment (interstitial or tissue fluid) and exert deleterious effects on cell functions. Much of this excess fluid collects relatively superficially within the skin, especially in the lower extremities or other dependent body parts as oedema.

The proposed study seeks to explore the possibility of significantly increasing the success rate (from the current rate of 28%) of clinically significant Transdermal Fluid Removal (TFR) in heart failure patients. It seeks to further understand the device and patient characteristics influencing successful clinically relevant fluid removal and to measure any patient-defined benefits. It also wishes to explore the patient experience of the removal.

Principal aim of the research: To investigate whether the TFR device can remove clinically viable or relevant volumes of fluid transdermally in advanced heart failure and other patients with significant oedema. "Clinically viable" volume is defined as the removal of 200ml or more of fluid in a session of up to 10 hours (or 0.43 ml/h per 1cm2 of the skin area treated with microneedles).

ELIGIBILITY:
Inclusion Criteria:

* Participants aged >18 years
* Diagnosis of heart failure
* Presence of visible oedema

Exclusion Criteria:

* Inability to give consent
* Patient on warfarin or simthrome (acecoumarol) with International Normalised Ratio (INR) >3 or other bleeding disorders
* Extensive skin disease, infected or broken skin over intended study area
* Pregnancy NB: Patients with pacemakers or implantable cardiac devices (ICD) may be recruited but will not have bioimpedance measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
Overall Success rate (volume): the % of patients that achieved the removal >200ml of fluid transdermally in a session. | 12 months
  Primary outcome/endpoint

SECONDARY OUTCOMES:
Overall Success rate (flow rate): % of patients in whom >0.43 ml/h per 1cm2 was removed using either 550µm or 850µm microneedles | 12 months
  % of patients in whom >0.43 ml/h per 1cm2 was removed using either 550µm or 850µm microneedles as reported on CRF
Success rate with short (550µm) and long (850 µm) microneedles respectively: % of patients in each category in whom >200ml or >0.43 ml/h per 1cm2 was removed | 12 months
  % of patients in each category in whom >200ml or >0.43 ml/h per 1cm2 was removed as reported on CRF
Microneedle insertion depth/force ratio: Mean (+SD) of microneedle skin insertion depth/insertion force used per microneedle type (550 µm and 850µm) | 12 months
  Mean (+SD) of microneedle skin insertion depth/insertion force used per microneedle type (550 µm and 850µm) as reported on CRF v1.0 and then analysed using appropriate statistics
Proportion of successfully penetration of microneedles per array: Tertile bands of successfully penetrated microneedle per array | 12 months
  Tertile bands of successfully penetrated microneedle per array
Incidence (%) of adverse rate per event and for all events | 12 months
  Adverse event rate: Incidence (%) of adverse rate per event and for all events as reported on AE log v4.0
Tolerability of TFR: N (%) in categories: "Well, very well, poorly or very poorly" tolerated. | 12 months
  N (%) in categories: "Well, very well, poorly or very poorly" tolerated reported on CRF
Characteristics of patients with successful versus unsuccessful TFR (e.g. demographics, extent of oedema, bioimpedance volumes, serum albumin) | 12 months
  N/mean/median (%/SD/IQR) as appropriate for single and multiple characteristics for "successful" and unsuccessful TFR groups as reported on CRF and then analysed using appropriate statistics.
Impact of the fluid extraction on routine activities including mobility, comfort, recovery experience: N (%) patients reporting "improved, no change or worsening" of each parameter. | 12 months
  N (%) patients reporting "improved, no change or worsening" of each parameter as reported on CRF, free text narrative and then analysed using appropriate statistics.
Patient' views on impact, usability and potential of the TFR device: N (%) patients reporting positive, negative or neutral in each category. | 12 months
  N (%) patients reporting positive, negative or neutral in each category, qualitative analysis and then analysed using appropriate statistics.

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom